CLINICAL TRIAL: NCT04443517
Title: EEG-Guided Analgesic Titration During General Anesthesia to Improve Early Neurocognitive Recovery in Older Patients
Acronym: ALPHA-DEX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Paul Garcia, Associate Professor of Anesthesiology, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAS4614
Record Dates: First submitted 2020-02-24; First posted 2020-06-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Delirium
Keywords: EEG; General Anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Maintenance-Alpha Optimization / Wake from Dexmedetomidine (Experimental): During the first randomization, participants randomized to intraoperative oscillatory EEG alpha optimization will receive individualized titration of anesthetic gas and opioids.
  Interventions: Procedure: Alpha Optimization; Behavioral: Emergence from anesthesia with Dexmedetomidine
- Maintenance-Alpha Optimization / Wake from Sevoflurane (Active Comparator): During the first randomization, participants randomized to intraoperative oscillatory EEG alpha optimization will receive real-time monitoring of alpha recordings and individualized titration of desflurane and opioid. During the second randomization, participants randomized to standard emergence from volatile anesthesia will be woken up per standard practice.
  Interventions: Procedure: Alpha Optimization
- Maintenance-Routine Care / Wake from Dexmedetomidine (Active Comparator): During the first randomization, participants randomized to standard of care will receive anesthesia per usual care with quantitative processed EEG index values and EEG wave forms.
  Interventions: Behavioral: Emergence from anesthesia with Dexmedetomidine
- Maintenance-Routine Care / Wake from Sevoflurane (No Intervention): During the first randomization, participants randomized to standard of care will receive anesthesia per usual care with quantitative processed EEG index values and EEG wave forms. During the second randomization, participants randomized to standard emergence from volatile anesthesia will be woken up per standard practice.

INTERVENTIONS:
Procedure: Alpha Optimization — Intraoperative oscillatory EEG alpha optimization involves real-time acquisition of oscillatory alpha power from the frontal EEG with individualized titration of sevoflurane and opioid.
  Arms: Maintenance-Alpha Optimization / Wake from Dexmedetomidine; Maintenance-Alpha Optimization / Wake from Sevoflurane
Behavioral: Emergence from anesthesia with Dexmedetomidine — Infusion of .05 mcg/kg/h of propofol during the final 10-20 minutes of surgery.
  Arms: Maintenance-Alpha Optimization / Wake from Dexmedetomidine; Maintenance-Routine Care / Wake from Dexmedetomidine

SUMMARY:
The investigators intend to recruit 600 participants to see if alpha power during anesthesia is influenced by analgesic medication and associated with a reduction of delirium following surgery.

DETAILED DESCRIPTION:
Postoperative delirium may manifest in the immediate post-anesthesia care period. Such episodes appear to be predictive of further episodes of inpatient delirium and associated adverse outcomes. Intraoperative monitoring of frontal electroencephalogram (EEG) has been associated with postoperative delirium and poor outcomes. However, the efficacy of titrating anesthesia medication to proprietary index targets for preventing delirium remains contentious. The investigators aim to assess the efficacy of two pharmacologic strategies which could prevent post-anesthesia care unit (PACU) delirium (1) maximization of intraoperative alpha power during maintenance and (2) switching anesthesia regimes during the emergence phases of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years or over
* Has capacity to provide informed consent
* Undergoing elective non-cardiac surgery, which does not involve the head or neck, with planned volatile-based general anesthesia of expected duration of at least 2 hours

Exclusion Criteria:

* Chronic pain with opioid requirement or concurrent use of enzyme inducers, e.g. carbamazepine, phenytoin,
* Illicit substance use or excessive alcohol intake
* Refusal by patient or case anesthesiologist responsible for patient's care

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Frontal Alpha Power | Up to 24 hours post-surgery
  The EEG data collected during the study duration will be processed using a customized script. Frontal alpha power (i.e., the cumulative power in the EEG alpha range) will be extracted from the EEGs and analyzed to compare the groups for the differences in the frontal alpha power.

SECONDARY OUTCOMES:
Incidence of PACU Delirium | Up to 24 hours post-surgery
  3-Minute Diagnostic Interview for Confusion Assessment Method(3D-CAM), Confusion Assessment Method for the ICU (CAM-ICU), Speech / Language Assessment will be administered to check for signs of delirium.
Change in pain in PACU: numerical rating score (NRS) | Up to 24 hours post-surgery
  The numerical rating score (NRS) requires the patient to rate their pain from 0-10 where 0 is no pain and 10 is the worst pain imaginable (high score indicates worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Garcia, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No